CLINICAL TRIAL: NCT01740765
Title: Energy Expenditure and Substrate Utilization During Acute Under- and Over-feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12-0681
Record Dates: First submitted 2012-11-18; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Energy Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eucaloric Feeding (Experimental): Subjects will complete an initial eucaloric feeding study day. During this study day, subjects will receive 100% of their calorie requirements. 24-hour energy expenditure will be measured.
  Interventions: Other: 24-hour energy expenditure
- Underfeeding (Experimental): Following the eucaloric feeding study day, subjects will undergo the underfeeding and overfeeding arms in random order. During the underfeeding study arm, subjects will receive 50% of their calorie requirements (as determined during the initial eucaloric study day) for 3 days. 24-hour energy expenditure will be measured.
  Interventions: Other: 24-hour energy expenditure
- Overfeeding (Experimental): Following the eucaloric feeding study day, subjects will undergo the underfeeding and overfeeding arms in random order. During the overfeeding study arm, subjects will receive 150% of their calorie requirements (as determined during the initial eucaloric study day) for 3 days. 24-hour energy expenditure will be measured.
  Interventions: Other: 24-hour energy expenditure

INTERVENTIONS:
Other: 24-hour energy expenditure — To assess 24-hour energy expenditure and substrate utilization subjects will spend 23 hours and 15 minutes each day in the metabolic chamber at the UNC NRI. Subjects will be requested to arrive at the study center each morning following a 10hour overnight fast. During each study day, subjects remained sedentary. All meals were provided and were tailored to each subject's specific energy requirements and the study protocol (i.e. 50% or 150% of calorie requirements).

SUMMARY:
This study will determine the impact of 24, 48 and 72 hours of over and underfeeding on energy expenditure as measured in the metabolic chamber at the UNC Chapel Hill Nutrition Research Institute (UNC NRI).

DETAILED DESCRIPTION:
Subjects will complete a baseline eucaloric study day. Following this, subjects will be randomized to complete 3 days of overfeeding (150% of baseline eucaloric energy requirements) or 3 days of underfeeding (50% of baseline eucaloric energy requirements). After completing one of these study arms, subjects will cross-over and complete the second arm. All study arms will be separated by two weeks. 24-hour energy expenditure will be measured 3 times during each of 3 day periods. We hypothesize that the impact of over or underfeeding on EE will be evident after 24-hours and will be comparable to 72 hour EE.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Postmenopausal
* Aged 50-65 years
* BMI 25-35kg/m2
* Not taking blood pressure or anti-inflammatory medications or any other medications that may impact the results
* Thyroid hormone profile within the normal reference range
* No medical condition which may impact the results (e.g. diabetes)
* Accustomed to eating regular meals including breakfast

Exclusion Criteria:

* Smoker
* Heavy exerciser (defined as >150 minutes/week for more than 3 months)
* Abuses alcohol or drugs
* Vegetarian

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure | 24-hour energy expenditure will be assessed
  24-hour energy expenditure will be assessed using the metabolic chamber at UNC NRI. Energy expenditure will be measured during eucaloric feeding (subjects will receive 100% of calorie requirements), as well as during 24, 48 and 72 hours of under and overfeeding.

SECONDARY OUTCOMES:
Whole blood transcriptomics | Fasting a.m. sample, before lunch, and at 0.5, 2, and 4.5 hours post lunch
  RNA will be extracted from whole blood. Transcriptomic profile will be assessed by microarray
Plasma metabolomics | Fasting a.m. sample, before lunch, and at 0.5, 2, and 4.5 hours post lunch
  Plasma metabolomic profile will be assessed using GC/MS and LC/MS platforms.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Swick, PhD, Principal Investigator — UNC Chapel Hill Nutrition Research Institute
Locations (1):
- UNC Chapel Hill Nutrition Research Institute, Kannapolis, North Carolina, United States